CLINICAL TRIAL: NCT06640244
Title: A Clinical Study to Evaluate the Efficacy of Prototypes for Improvement in Skin Tone and Spot Brightening in a Full-Face Study Design
Brief Title: The Effect of Cosmetic Face Care Products on Facial Skin Tone and Spot Brightening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: MS Clinical Research Pvt. Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMN-SKA-4185
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pigment Spots
MeSH Terms: interventions — Sunscreening Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cosmetic product G18 (Experimental): Cosmetic face care product to be used twice daily on the whole face for 12 weeks.
  Interventions: Other: Sunscreen; Other: Cosmetic product G18
- Cosmetic product N70 (Experimental): Cosmetic face care product to be used twice daily on the whole face for 12 weeks.
  Interventions: Other: Sunscreen; Other: Cosmetic product N70
- Cosmetic product D79 (Experimental): Cosmetic face care product to be used twice daily on the whole face for 12 weeks.
  Interventions: Other: Sunscreen; Other: Cosmetic product D79
- Cosmetic product E84 (Experimental): Cosmetic face care product to be used twice daily on the whole face for 12 weeks.
  Interventions: Other: Sunscreen; Other: Cosmetic product E84
- Cosmetic product C68 (Experimental): Cosmetic face care product to be used twice daily on the whole face for 12 weeks.
  Interventions: Other: Sunscreen; Other: Cosmetic product C68

INTERVENTIONS:
Other: Sunscreen — To be used by all participants throughout the study
Other: Cosmetic product G18 — Cosmetic face care product
  Arms: Cosmetic product G18
Other: Cosmetic product N70 — Cosmetic face care product
  Arms: Cosmetic product N70
Other: Cosmetic product D79 — Cosmetic face care product
  Arms: Cosmetic product D79
Other: Cosmetic product E84 — Cosmetic face care product
  Arms: Cosmetic product E84
Other: Cosmetic product C68 — Cosmetic face care product
  Arms: Cosmetic product C68

SUMMARY:
This is a single centre, 5-cell, blinded study to evaluate changes in even skin tone, skin glow, facial pigmented spots, and the microbiome of facial skin following the use of cosmetic face care products on the whole face over a 12 week period.

DETAILED DESCRIPTION:
This is a randomized, blinded, 5 cell, full-face study designed to evaluate changes in even skin tone, skin glow, pigmented spots and the surface microbiome of facial skin following the use of one of five cosmetic face care products. This study will accept up to 50 participants per cell (250 participants overall) who meet the inclusion/exclusion criteria to ensure that at least 40 participants per cell complete the study. Participants will be randomised to receive one of the five cosmetic face care products which will be applied to the whole face using a defined protocol.

If accepted onto the study, all participants will be provided with a marketed face wash to use for one week prior to the baseline visit and throughout the whole study.

Visual and instrumental assessments of skin colour, skin glow and even tone will be conducted throughout the duration of the study (12 weeks product use and 6 weeks regression). Non-invasive skin surface samples will be collected at several timepoints for evaluation of the skin microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Female adult participants in general good health as determined from a recent medical history.
* Participants in the age group of 20-45 years (both ages inclusive).
* Participants having Fitzpatrick photo-type III-V.
* Participants with at least 3 spots on the cheek either of PIH post acne/age related
* Participants not presenting any skin condition that may interfere with the assessment for the entire study duration.
* Participants free of excessive hair, acne, cuts, abrasions, fissures, wounds, lacerations, or any other active skin conditions on the face
* Participant who agrees not to use any other product/treatment/home remedy/serum on their face during the study period other than the study product.
* Participants who agree to remove all jewellery on/around face (e.g., necklace, earrings, nose ring), during imaging.
* Participants willing to give a voluntary written informed consent and photography release.
* Participants willing to abide by and comply with the study protocol.
* Participants able to read, understand and sign an appropriate informed consent form indicating her willingness to participate.
* Participants willing and capable to follow the study rules and a fixed schedule.

Exclusion Criteria:

* Participants who are currently participating in a similar study or have participated in a similar study in the past 6 weeks.
* Participants with any other signs of significant local irritation, erythema, or skin disease on skin.
* Participants having chronic illness or who have undergone major surgery in the last year that may be clinically relevant or can impact the results as determined by the dermatologist.
* Participants undergoing treatment for any skin condition.
* Participants allergic or sensitive to bar cleansing products, creams/lotions, artificial jewellery or anything else.
* Participants with self-perceived pimple prone and/or sensitive skin.
* Participants taking any oral antibiotic medication currently or within the last 8 weeks.
* Participants taking medication continuously/regularly every day such as corticosteroids or non-steroidal anti-inflammatories, topically for four weeks or orally for eight weeks prior to the study.
* Female participant pregnant/breast feeding or planning pregnancy during the study period (self-declared)
* Participants taking product/treatment for any condition which the Investigator believes may influence the interpretation of the data.
* Participants currently taking any medication, which the investigator believes may influence the interpretation of the data.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Visual assessment of skin colour | 0-12 weeks + 6 weeks regression
Instrumental assessment of skin colour | 0-12 weeks + 6 weeks regression

SECONDARY OUTCOMES:
Changes in skin surface microbiome | 0-12 weeks + 6 weeks regression

OTHER OUTCOMES:
Self assessment questionnaires | 0-12 weeks + 6 weeks regression
Visual assessment of facial skin glow and radiance. | 0-12 weeks + 6 weeks regression

CONTACTS AND LOCATIONS:
Locations (1):
- MS Clinical Research Pvt Ltd, Bangalore, India

IPD SHARING:
Plan to Share IPD: No